CLINICAL TRIAL: NCT01659541
Title: Spinal Cord Stimulation With Wire Leads to Restore Cough
Brief Title: Stimulation With Wire Leads to Restore Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Anthony F. Dimarco, Professor, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 15-00014; U01NS083696 (NIH)
Record Dates: First submitted 2012-05-23; First posted 2012-08-08 (Estimated); Results first posted 2022-08-19 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases; Paralysis; Central Nervous System Diseases; Cough; Trauma, Nervous System; Wounds and Injuries
Keywords: spinal cord injury; paralysis; cough; cervical spinal cord injury; thoracic spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases; Paralysis; Central Nervous System Diseases; Cough; Trauma, Nervous System; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Procedure & Device (Experimental): Procedure/Surgery: Implantation of device; Device: Expiratory Muscle Stimulator
  Interventions: Device: Expiratory muscle stimulator; Procedure: Implantation of device

INTERVENTIONS:
Device: Expiratory muscle stimulator — The expiratory muscle stimulator consists of two small electrodes (wire leads) implanted on the surface of the spinal cord on the lower back to stimulate the expiratory muscles and restore cough. These electrodes are connected to an implanted receiver in the abdomen or chest wall. The device is activated through an external antenna connected to an external control box.
  Other Names: Custom Finetech/Ardiem Sacral Anterior Root Stimulator
Procedure: Implantation of device — The expiratory muscle stimulator consists of two wire leads(each with two metal contacts) inserted onto the surface of their spinal cord on the lower back using a needle. The procedure to implant these wire leads is commonly used today for other purposes. This is a minimally invasive surgical technique with minimal risks. The wire leads are connected to an implanted receiver in the abdomen or chest wall. The device is activated through an external antenna connected to an external control box to stimulate the expiratory muscles and restore cough.

SUMMARY:
The purpose of this trial is to determine the efficacy of spinal cord stimulation, using wire leads, to produce an effective cough in patients with spinal cord injuries.

DETAILED DESCRIPTION:
Patients with cervical spinal cord injuries often have paralysis of a major portion of their expiratory muscles - the muscles responsible for coughing - and therefore, lack a normal cough mechanism. Consequently, most of these patients suffer from a markedly reduced ability to clear airway secretions, a factor which contributes to the development of recurrent respiratory tract infections such as pneumonia and bronchitis. Expiratory muscles can be activated by electrical stimulation of the spinal roots to produce a functionally effective cough.

The purpose of this trial is to determine if electrical stimulation of the expiratory muscles by wire leads is capable of producing an effective cough on demand. According to the trial researchers, if successful, this technique will prevent the need for frequent patient suctioning - which often requires the constant presence of trained personnel. It will also allow spinal cord injured patients to clear their secretions more readily, thereby reducing the incidence of respiratory complications and associated illness and death.

In the trial, researchers will study 16 adults (18-75 years old) with cervical spinal injuries (C8 level or higher), at least 6 months following the date of injury. After an evaluation of medical history, a brief physical examination, and initial testing, participants will have wire leads placed - by a routine, minimally invasive surgical procedure - over the surface of their spinal cords on the lower back to stimulate the expiratory muscles and restore cough.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury C8 level or higher
* 12 months post-injury (if the American Spinal Injury Association (ASIA) Impairment Scale (AIS) incomplete) or 6 months post-injury (if AIS complete)
* Expiratory muscle weakness
* Between 18 and 75 years of age
* Adequate oxygenation

Exclusion Criteria:

* Untreated lung, cardiovascular or brain disease
* Scoliosis, chest wall deformity, or marked obesity
* Unmanaged hypertension (high blood pressure) or hypotension (low blood pressure)
* Low oxygenation
* Minor infection at the site of implantation requiring antibiotics within the past 3 weeks
* Serious infection requiring hospitalization within the past 6 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F. DiMarco, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] DiMarco AF, Kowalski KE, Geertman RT, Hromyak DR. Spinal cord stimulation: a new method to produce an effective cough in patients with spinal cord injury. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1386-9. doi: 10.1164/rccm.200601-097CR. Epub 2006 Mar 16. PMID 16543552
- [Background] DiMarco AF, Kowalski KE, Geertman RT, Hromyak DR, Frost FS, Creasey GH, Nemunaitis GA. Lower thoracic spinal cord stimulation to restore cough in patients with spinal cord injury: results of a National Institutes of Health-Sponsored clinical trial. Part II: clinical outcomes. Arch Phys Med Rehabil. 2009 May;90(5):726-32. doi: 10.1016/j.apmr.2008.11.014. PMID 19406290
- [Background] DiMarco AF, Kowalski KE, Geertman RT, Hromyak DR. Lower thoracic spinal cord stimulation to restore cough in patients with spinal cord injury: results of a National Institutes of Health-sponsored clinical trial. Part I: methodology and effectiveness of expiratory muscle activation. Arch Phys Med Rehabil. 2009 May;90(5):717-25. doi: 10.1016/j.apmr.2008.11.013. PMID 19406289
- [Background] Kowalski KE, DiMarco AF. Comparison of wire and disc leads to activate the expiratory muscles in dogs. J Spinal Cord Med. 2011 Nov;34(6):600-8. doi: 10.1179/2045772311Y.0000000039. PMID 22330116
- [Background] DiMarco AF, Romaniuk JR, Supinski GS. Electrical activation of the expiratory muscles to restore cough. Am J Respir Crit Care Med. 1995 May;151(5):1466-71. doi: 10.1164/ajrccm.151.5.7735601.
- [Background] DiMarco AF, Romaniuk JR, Kowalski KE, Supinski G. Pattern of expiratory muscle activation during lower thoracic spinal cord stimulation. J Appl Physiol (1985). 1999 Jun;86(6):1881-9. doi: 10.1152/jappl.1999.86.6.1881. PMID 10368352
- [Background] DiMarco AF, Romaniuk JR, Kowalski KE, Supinski G. Mechanical contribution of expiratory muscles to pressure generation during spinal cord stimulation. J Appl Physiol (1985). 1999 Oct;87(4):1433-9. doi: 10.1152/jappl.1999.87.4.1433. PMID 10517775
- [Background] Wada JA, Osawa T, Mizoguchi T. Recurrent spontaneous seizure state induced by prefrontal kindling in senegalese baboons, Papio papio. Can J Neurol Sci. 1975 Nov;2(4):477-92. doi: 10.1017/s031716710002062x. PMID 1201534
- [Background] Romaniuk JR, Dick TE, Kowalski KE, Dimarco AF. Effects of pulse lung inflation on chest wall expiratory motor activity. J Appl Physiol (1985). 2007 Jan;102(1):485-91. doi: 10.1152/japplphysiol.00130.2006. Epub 2006 Sep 7. PMID 16959914
- [Background] Kowalski KE, Romaniuk JR, DiMarco AF. Changes in expiratory muscle function following spinal cord section. J Appl Physiol (1985). 2007 Apr;102(4):1422-8. doi: 10.1152/japplphysiol.00870.2006. Epub 2006 Dec 7. PMID 17158247
- [Background] DiMarco AF, Kowalski KE, Romaniuk JR. Effects of diaphragm activation on airway pressure generation during lower thoracic spinal cord stimulation. Respir Physiol Neurobiol. 2007 Oct 15;159(1):102-7. doi: 10.1016/j.resp.2007.06.007. Epub 2007 Jun 22. PMID 17681870
- [Background] DiMarco AF, Kowalski KE. Effects of chronic electrical stimulation on paralyzed expiratory muscles. J Appl Physiol (1985). 2008 Jun;104(6):1634-40. doi: 10.1152/japplphysiol.01321.2007. Epub 2008 Apr 10. PMID 18403449
- [Background] DiMarco AF, Kowalski KE, Hromyak DR, Geertman RT. Long-term follow-up of spinal cord stimulation to restore cough in subjects with spinal cord injury. J Spinal Cord Med. 2014 Jul;37(4):380-8. doi: 10.1179/2045772313Y.0000000152. Epub 2013 Nov 26. PMID 24090524
- [Background] DiMarco AF, Geertman RT, Tabbaa K, Polito RR, Kowalski KE. Economic Consequences of an Implanted Neuroprosthesis in Subjects with Spinal Cord Injury for Restoration of an Effective Cough. Top Spinal Cord Inj Rehabil. 2017 Summer;23(3):271-278. doi: 10.1310/sci2303-271. PMID 29339903
- [Background] DiMarco AF, Geertman RT, Tabbaa K, Polito RR, Kowalski KE. Case report: Minimally invasive method to activate the expiratory muscles to restore cough. J Spinal Cord Med. 2018 Sep;41(5):562-566. doi: 10.1080/10790268.2017.1357916. Epub 2017 Oct 11. PMID 29017400
- [Background] DiMarco AF, Geertman RT, Tabbaa K, Kowalski KE. Complete Restoration of Respiratory Muscle Function in Three Subjects With Spinal Cord Injury: Pilot Interventional Clinical Trial. Am J Phys Med Rehabil. 2019 Jan;98(1):43-50. doi: 10.1097/PHM.0000000000001018. PMID 30119089
- [Background] DiMarco AF, Geertman RT, Tabbaa K, Nemunaitis GA and Kowalski KE. Case Report: Effects of Lower Thoracic Spinal Cord Stimulation on Bowel Management in a Person with Spinal Cord Injury. Journal of Neurology and Neurobiology (2019) Volume 5 - Issue 1 | DOI: http://dx.doi.org/10.16966/2379-7150.156.
- [Background] DiMarco AF, Geertman RT, Tabbaa K, Kowalski KE. Complete Restoration of Respiratory Muscle Function in Subjects With Spinal Cord Injury: Interventional Clinical Trial. Am J Phys Med Rehabil. 2020 Jul;99(7):e91-e92. doi: 10.1097/PHM.0000000000001338. No abstract available. PMID 31688014
- [Background] DiMarco AF, Geertman RT, Tabbaa K, Nemunaitis GA, Kowalski KE. Restoration of cough via spinal cord stimulation improves pulmonary function in tetraplegics. J Spinal Cord Med. 2020 Sep;43(5):579-585. doi: 10.1080/10790268.2019.1699678. Epub 2019 Dec 6. PMID 31809251
- [Background] DiMarco AF, Geertman RT, Tabbaa K, Nemunaitis GA, Kowalski KE. Effects of Lower Thoracic Spinal Cord Stimulation on Bowel Management in Individuals With Spinal Cord Injury. Arch Phys Med Rehabil. 2021 Jun;102(6):1155-1164. doi: 10.1016/j.apmr.2020.09.394. Epub 2020 Nov 5. PMID 33161007
- [Background] DiMarco AF, Geertman RT, Nemunaitis GA, Kowalski KE. Comparison of disc and wire electrodes to restore cough via lower thoracic spinal cord stimulation. J Spinal Cord Med. 2022 May;45(3):354-363. doi: 10.1080/10790268.2021.1936388. Epub 2021 Jul 7. PMID 34232841
- [Derived] DiMarco AF, Geertman RT, Nemunaitis GA, Kowalski KE. Impact of the cough stimulation system on the care burden and life quality of caregivers of tetraplegics. J Spinal Cord Med. 2023 Sep;46(5):778-788. doi: 10.1080/10790268.2022.2148845. Epub 2023 Apr 5. PMID 37017634

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were well informed of the details of the study, with particular interest to risks/benefits, and asked to review the Informed Consent before signing. They were given an opportunity to ask questions. Consent was obtained only after all questions and concerns have been addressed.
Groups:
- Spinal Cord Stimulation With Wire Leads to Restore Cough: Procedure/Surgery: Implantation of device; Device: Expiratory Muscle Stimulator
  Expiratory muscle stimulator: The expiratory muscle stimulator consists of two small electrodes (wire leads) implanted on the surface of the spinal cord on the lower back to stimulate the expiratory muscles and restore cough. These electrodes are connected to an implanted receiver in the abdomen or chest wall. The device is activated through an external antenna connected to an external control box.
  Implantation of device: The expiratory muscle stimulator consists of two wire leads(each with two metal contacts) inserted onto the surface of their spinal cord on the lower back using a needle. The procedure to implant these wire leads is commonly used today for other purposes. This is a minimally invasive surgical technique with minimal risks. The wire leads are connected to an implanted receiver in the abdomen or chest wall. The device is activated through an external antenna connected to an external control box to stimulate the expiratory muscles and restore cough.
Period: Overall Study
Arm/Group | Spinal Cord Stimulation With Wire Leads to Restore Cough
Started | 12
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Clinical Trial: Spinal Cord Stimulation to Restore Cough: Procedure/Surgery: Implantation of device; Device: Expiratory Muscle Stimulator
  Expiratory muscle stimulator: The expiratory muscle stimulator consists of two small electrodes (wire leads) implanted on the surface of the spinal cord on the lower back to stimulate the expiratory muscles and restore cough. These electrodes are connected to an implanted receiver in the abdomen or chest wall. The device is activated through an external antenna connected to an external control box.
  Implantation of device: The expiratory muscle stimulator consists of two wire leads(each with two metal contacts) inserted onto the surface of their spinal cord on the lower back using a needle. The procedure to implant these wire leads is commonly used today for other purposes. This is a minimally invasive surgical technique with minimal risks. The wire leads are connected to an implanted receiver in the abdomen or chest wall. The device is activated through an external antenna connected to an external control box to stimulate the expiratory muscles and restore cough.
Arm/Group | Clinical Trial: Spinal Cord Stimulation to Restore Cough
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12
Region of Enrollment [Number; unit: participants]
  United States | 12
Pre-Implant - Spontaneous Effort - Airway Pressure [Mean (Standard Deviation); unit: cmH2O] — Population: A medical implant (cough system) has been removed (explanted ) from one participant due to increase in frequency and severity of spasms.
  cmH2O
    number analyzed (Participants) | 11
    (all) | 24.7 (12.9)

OUTCOME MEASURES:

1. Primary Outcome: Measurements of Peak Expiratory Airflow Rate to Evaluate Efficacy of Cough.
Description: Peak Expiratory airflow rate is a person's maximum speed of expiration. Peak expiratory flow rate is the maximum flow rate generated during a forceful exhalation, starting from full inspiration. It was measured after release of airway occlusion after peak airway pressure was achieved.
Time Frame: 52 weeks (1 year)
Measure: Mean (Standard Error); unit: L/s
Groups:
- Peak Expiratory Airflow Rate (L/s): Each patient was served as their own control (Pre-Implant); comparisons were made at various points in the study (Week #28, #40 and #52).
Arm/Group | Peak Expiratory Airflow Rate (L/s)
Number analyzed (Participants) | 11
L/s
  Pre-Implant - Spontaneous Effort | 2.1 (0.4)
  Post-Implantation Week #28 | 9.6 (1.2)
  Post-Implantation Week #40 | 10.4 (1.3)
  Post-Implantation Week #52 | 11.1 (1.6)
Statistical Analysis 1: Comparison: Peak Expiratory Airflow Rate (L/s); Each patient was served as their own control (Pre-Implant); comparisons was made at various points in the study (Week #28, #40 and #52); Test type: Other — Statistical analyses were performed using a repeated measures analysis of variance and Paired t test. A p value was calculated; p < 0.05, ANOVA; Statistical analyses will be performed using a repeated measures analysis of variance and Paired t test

2. Primary Outcome: Measurements of Maximum Airway Pressure to Evaluate Efficacy of Cough
Description: Maximum expiratory pressure is the highest pressure that can be developed during a forceful expiratory effort against an occluded airway.
Time Frame: 52 weeks (1 year)
Measure: Mean (Standard Error); unit: cmH2O
Groups:
- Maximum Airway Pressure Generation: Airway pressure generation measurements were made under conditions of airway occlusion during subject spontaneous effort and during spinal cord stimulation (Cough System) at total lung capacity (TLC) with subject maximal expiratory effort.
  Each patient was served as their own control (Pre-Implant); comparisons were made at various points in the study (Week #28, #40 and #52).
Arm/Group | Maximum Airway Pressure Generation
Number analyzed (Participants) | 11
cmH2O
  Pre-Implant -Spontaneous Effort | 25 (4)
  Post-Implantation Week #28 | 112 (13)
  Post-Implantation Week #40 | 117 (14)
  Post-Implantation Week #52 | 118 (14)
Statistical Analysis 1: Comparison: Maximum Airway Pressure Generation; Each patient was served as their own control (Pre-Implant); comparisons were made at various points in the study (Week #28, #40 and #52); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA; Statistical analyses will be performed using a repeated measures analysis of variance and Paired t test

3. Secondary Outcome: Secretion Management Episodes
Description: This assessment allowed to characterize the severity of secretion management episodes and subjective assessment of the need for secretion management before and after use of the Cough System.
  Design: Prospective assessment via questionnaire responses
  Question: How significant were your needs for assistance with managing your airway secretions on a typical day during the past week?
  0 None - Unaware of need
  1. Mild - Did not interfere with usual daily activities
  2. Moderate - Most stop activity during need
  3. Marked - Most stop activity for brief period (10-30 min) after need
  4. Severe - Most stop activity for prolonged period (> 30 min) after need, may be accompanied by dizziness, headache and/or pain in upper chest
Time Frame: 52 weeks (1 year)
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Secretion Management Episodes: This assessment allowed to characterize the severity of secretion management episodes and subjective assessment of the need for secretion management before (Pre-Implant) and after use of the Cough System.
  Design: Prospective assessment via questionnaire responses
  Question: How significant were your needs for assistance with managing your airway secretions on a typical day during the past week?
  0 None - Unaware of need
  1. Mild - Did not interfere with usual daily activities
  2. Moderate - Most stop activity during need
  3. Marked - Most stop activity for brief period (10-30 min) after need
  4. Severe - Most stop activity for prolonged period (> 30 min) after need, may be accompanied by dizziness, headache and/or pain in upper chest
  Each patient was served as their own control (Pre-Implant); comparisons were made at various points in the study (Week #28, #40 and #52).
Arm/Group | Secretion Management Episodes
Number analyzed (Participants) | 11
score on a scale
  Pre-Implant | 2.73 (0.41)
  Post-Implantation Week #28 | 0.45 (0.21)
  Post-Implantation Week #40 | 0.55 (0.21)
  Post-Implantation Week #52 | 0.45 (0.21)
Statistical Analysis 1: Comparison: Secretion Management Episodes; The data prior to implantation (Pre-Implant)) were compared with data obtained after implantation (Week ##28, #40, #52) of the cough system using a nonparametric analog (Friedman Test) to the standard repeated measures analysis of variance. A p value was calculated. This alpha level was chosen as a correlation for inflated type I error rates because of multiple comparisons. Results are reported as means ± Standard Error; Test type: Other; p < 0.05, nonparametric analog (Freidman Test)

4. Secondary Outcome: Difficulty Raising Sputum
Description: Survey to assess difficulty raising sputum
  Objectives: To determine the difficulty raising sputum before and after use of the cough stimulation system (Cough System)
  Design: Prospective assessment via questionnaire responses
  Question: How much difficulty have you had with managing your airway secretions?
  On a scale of 0-4 (0 = None (No secretions), 1 = Mild (Rarely have difficulty), 2 = Moderate (Occasional difficulty) 3 = Marked (Frequent difficulty) and 4=Severe (Usually have great difficulty).
Time Frame: 52 weeks (1 year)
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Difficulty Raising Sputum: Survey to assess difficulty raising sputum
  Objectives: To determine the difficulty raising sputum before (Pre-Implant) and after use of the cough stimulation system (Cough System)
  Design: Prospective assessment via questionnaire responses
  Question: How much difficulty have you had with managing your airway secretions?
  On a scale of 0-4 (0 = None (No secretions), 1 = Mild (Rarely have difficulty), 2 = Moderate (Occasional difficulty) 3 = Marked (Frequent difficulty) and 4=Severe (Usually have great difficulty).
  Each patient was served as their own control (Pre-Implant); comparisons were made at various points in the study (Week #28, #40 and #52).
Arm/Group | Difficulty Raising Sputum
Number analyzed (Participants) | 11
score on a scale
  Pre-Implantation | 2.64 (0.41)
  Post-Implantation Week #28 | 0.64 (0.24)
  Post-Implantation Week #40 | 0.55 (0.21)
  Post-Implantation Week #52 | 0.36 (0.20)
Statistical Analysis 1: Comparison: Difficulty Raising Sputum; The data prior to implantation (Pre-Implant) were compared with data obtained after implantation (Week #28, #40, #52) of the cough system using a nonparametric analog (Friedman Test) to the standard repeated measures analysis of variance. A p value was calculated. This alpha level was chosen as a correlation for inflated type I error rates because of multiple comparisons. Results are reported as means ± Standard Error; Test type: Other; p < 0.05, nonparametric analog (Freidman Test)

5. Secondary Outcome: Number of Respiratory Tract Infections
Description: Form covers frequency, type, severity, and antibiotic use for respiratory tract infections.
  The incidence of acute respiratory tract infections, defined by a change in the character, color, or amount of respiratory secretions and requiring antibiotic administration was tracked before and after implantation of the cough system. The occurrence of respiratory tract infections was determined by subject history and corroborated by review of medical records, when available.
Time Frame: 52 weeks (1 year)
Measure: Mean (Standard Error); unit: Respiratory tract infections per year
Groups:
- Number of Respiratory Tract Infections: Pre-Implantation; Number of Respiratory Tract Infections: Post-Implant - After Use of the Cough System (Week #52): The incidence of acute respiratory tract infections, defined by a change in the character, color, or amount of respiratory secretions and requiring antibiotic administration was tracked before and after use of the Cough System.
  The occurrence of respiratory tract infections was determined by subject history and corroborated by review of medical records, when available.
Arm/Group | Number of Respiratory Tract Infections: Pre-Implantation | Number of Respiratory Tract Infections: Post-Implant - After Use of the Cough System (Week #52)
Number analyzed (Participants) | 11 | 11
Respiratory tract infections per year | 1.5 (0.6) | 0.1 (0.1)
Statistical Analysis 1: Comparison: Number of Respiratory Tract Infections: Pre-Implantation vs Number of Respiratory Tract Infections: Post-Implant - After Use of the Cough System (Week #52); The data prior to implantation (Pre-Implant) were compared with data obtained after implantation (Week #28 ,#40, #52) of the cough system using a nonparametric analog (Friedman Test) to the standard repeated measures analysis of variance. Paired t test. A p value was calculated. This alpha level was chosen as a correlation for inflated type I error rates because of multiple comparisons. Results are reported as means ± Standard Error; Test type: Other; p < 0.05, nonparametric analog (Freidman Test)

6. Secondary Outcome: Life Quality Assessment -Stress Level
Description: Survey will assess the subject's quality of life at home and in social situations, as well as assess specific need for managing secretions.
  Objectives: Life Quality Assessment before and after use of the cough stimulation system (Cough System)
  Design: Prospective assessment via questionnaire responses
  Question: To what extent did managing your airway secretions cause you stress? On a scale of 0-3 (0 = Not at all, 1 = a little, 2 = Quite a bit and 3 = Very much)
Time Frame: 52 weeks (1 year)
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Life Quality Assessment (Stress Level): Participant Life Quality Assessment: before (Pre-Implant) and after use of the cough stimulation system (Cough System)
  Design: Prospective assessment via questionnaire responses
  Question: To what extent did managing your airway secretions cause you stress? On a scale of 0-3 (0 = Not at all, 1 = a little, 2 = Quite a bit and 3 = Very much)
  Each patient was served as their own control (Pre-Implant); comparisons were made at various points in the study (Week #28, #40 and #52).
Arm/Group | Life Quality Assessment (Stress Level)
Number analyzed (Participants) | 11
score on a scale
  Pre-Implantation | 2.27 (0.24)
  Post-Implantation Week #28 | 0.18 (0.18)
  Post-Implantation Week #40 | 0.18 (0.18)
  Post-Implantation Week #52 | 0.27 (0.27)
Statistical Analysis 1: Comparison: Life Quality Assessment (Stress Level); [analysis description as in outcome 4, analysis 1]; Test type: Other; p < 0.05, nonparametric analog (Freidman Test)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Post-Implantation; Spinal Cord Stimulation With Wire Leads to Restore Cough: Procedure/Surgery: Implantation of device; Device: Expiratory Muscle Stimulator
  The expiratory muscle stimulator (Cough System) consists of two small electrodes (wire leads) implanted on the surface of the spinal cord on the lower back to stimulate the expiratory muscles and restore cough. These electrodes are connected to an implanted receiver in the abdomen or chest wall. The device is activated through an external antenna connected to an external control box.
  Use of the spinal cord stimulation (SCS) Cough System was associated with some side effects, most notably increases in blood pressure and decreases in heart rate, consistent with autonomic dysreflexia (AD). AD was limited to the early phase of SCS and occurred in a total of 6 subjects. Over a period of several weeks of daily SCS however, this response gradually abated and eventually resolved in each subject. Mild back and leg jerking without associated discomfort was also observed in some subjects. This effect was well controlled by reducing the intensity of SCS.
  There was no evidence of bowel or bladder leakage.
  The Cough System have had to be explanted in one participant due increase in frequency and severity of muscle spasm.
Arm/Group | Post-Implantation; Spinal Cord Stimulation With Wire Leads to Restore Cough
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-Implantation; Spinal Cord Stimulation With Wire Leads to Restore Cough (N=12)
Hemodynamic effect - Initial increases in blood pressure and decreases in heart rate (Nervous system disorders) | 6 (6) — Use of the Cough System was associated with some side effects (n=6), most notably increases in blood pressure, consistent with AD. Over a period of several weeks of daily SCS however, those responses were eventually resolved in each subject.
Muscle spasm (Nervous system disorders) | 1 (1) — The Cough System have had to be explanted in one participant due an increase in frequency and severity of muscle spasm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT01659541/Prot_000.pdf
  • Statistical Analysis Plan (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT01659541/SAP_001.pdf
  • Informed Consent Form (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT01659541/ICF_002.pdf